CLINICAL TRIAL: NCT03896451
Title: Prospactive Randomized Monocentric Comparison Study Between Two Total Knee Prosthesis Medacta GMK Sphere and Medacta GMK PS
Brief Title: Comparison Between Two Total Knee Prosthesis Medacta GMK Sphere and Medacta GMK PS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Medacta GMK PS is not in use anymore
Sponsor: Kantonsspital Winterthur KSW (Other)
Responsible Party: Principal Investigator, Peter Koch, Principal Investigator: PD/MD, Kantonsspital Winterthur KSW
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: PS vs. Sphere
Record Dates: First submitted 2019-03-26; First posted 2019-04-01 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GMK Sphere (Other): Patients receiving total knee replacement surgery with the device "Medacta GMK Sphere"
  Interventions: Device: Total knee endoprothesis
- GMK PS (Other): Patients receiving total knee replacement surgery with the device "Medacta GMK PS"
  Interventions: Device: Total knee endoprothesis

INTERVENTIONS:
Device: Total knee endoprothesis — Total knee endoprosthesis after knee joint osteoarthritis

SUMMARY:
The purpose of the study is to compare the clinical outcome after two total knee endoprosthesis designs Medacta GMK Sphere and Medacta GMK PS.

Primary outcome measures KOOS, Forgotten Knee Score and range of motion.

Single-center, randomized trial

DETAILED DESCRIPTION:
The clinical outcome measures were measured preoperativ and postoperativ (1 year, 5 year and 10 year).

Secondary outcome measures: number of reoperations and revisions, survival of the prosthesis

The patient population would consist patients with knee osteoarthritis eligible for total knee replacement

The aim of the study is to evaluate the effect of the knee prosthesis design on the patient outcome

ELIGIBILITY:
Inclusion Criteria:

* patient is eligible for a total knee replacement
* patient is eligible for a Medacta GMK Sphere or Medacta GMK PS knee prosthesis
* patient signed the informed consent

Exclusion Criteria:

* patient is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-02 (Actual); Primary Completion 2031-03-31 (Estimated); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Knee injury and Osteoarthritis Outcome Score | preoperative, 1 year, 5 year and 10 year after surgery
  Knee injury and Osteoarthritis Outcome Score: 100 = maximum score, 0 = minimum score
Change in Forgotten Joint Score | 1 year, 5 year and 10 year after surgery
  Forgotten Joint Score: 100 = maximum score, 0 = minimum score

SECONDARY OUTCOMES:
Change in revison | 1 year, 5 year and 10 year after surgery
  Revision rate comparision with the baseline at 1 year
Change in range of motion | preoperative, 1 year, 5 year and 10 year after surgery
  Range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Peter Koch, PD Dr. med., Principal Investigator — Principal Investigator
Locations (1):
- Kantonsspital Winterthur, Winterthur, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No